CLINICAL TRIAL: NCT05663476
Title: Effect Of Non Surgical Therapy On Vitronectin And Fetuin-A Levels In Patients With Periodontitis And Coronary Artery Disease- An Interventional Study
Brief Title: NSPT On Vitronectin And Fetuin-A Levels In Patients With Periodontitis And Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Director of Research, Meenakshi Ammal Dental College and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADC/IEC-1/18/2022
Record Dates: First submitted 2022-11-10; First posted 2022-12-23 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Chronic Periodontitis; Cardiovascular Diseases; Periodontal Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Three arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Periodontally and systemically healthy participants
  Interventions: Other: Non Surgical Periodontal Therapy
- Periodontitis without coronary artery disease (Experimental): Periodontitis participants without coronary artery disease
  Interventions: Other: Non Surgical Periodontal Therapy
- Periodontitis with coronary artery disease (Experimental): Periodontitis participants with coronary artery disease
  Interventions: Other: Non Surgical Periodontal Therapy

INTERVENTIONS:
Other: Non Surgical Periodontal Therapy — Scaling and root planing using scalers and periodontal curettes will be done

SUMMARY:
Periodontitis is a chronic inflammatory disease mainly caused by the oral microbial biofilm. It involves the periodontal supporting tissues mainly features gum inflammation, alveolar bone resorption, periodontal pocket formation, and tooth loosening but also induces various systemic diseases, which seriously affect the physical and mental health of patients. The response to periodontal infection is mediated by various intracellular signalling pathways leading to the production of numerous bio-molecules. Vitronectin is a multifunctional protein with a multiple binding domain that interacts with a variety of plasma and cell proteins. It belongs to the group of adhesive glycoproteins that is involved in various functions including complement activation, blood coagulation, binding to proteoglycans, and modification of the matrix. Among the various cystatins expressed in serum and saliva, Fetuin-A, an another protein is produced majorly by healthy hepatic and adipose tissues. Fetuin-A has been recognized as a multifunctional molecule related to its role in metabolic processes, insulin resistance, regulation of adipogenesis and mineralization throughout the body. The study aims to determine the expression of Vitronectin and Fetuin-A as potential pro-inflammatory and anti-inflammatory biomarkers respectively. These protein molecules can further play a role as putative risk indicators in periodontitis subjects with and without coronary artery disease following non-surgical therapy.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease mainly caused by the oral microbial biofilm. It involves the periodontal supporting tissues mainly features gum inflammation, alveolar bone resorption, periodontal pocket formation, and tooth loosening but also induces various systemic diseases, which seriously affect the physical and mental health of patients. The response to periodontal infection is mediated by various intracellular signaling pathways leading to the production of numerous bio-molecules. Vitronectin is a multifunctional protein with multiple binding domains that interact with a variety of plasma and cell proteins. It belongs to the group of adhesive glycoproteins that are involved in various functions including complement activation, blood coagulation, binding to proteoglycans, and modification of the matrix. Among the various cystatins expressed in serum and saliva, Fetuin-A, another protein is produced majorly by healthy hepatic and adipose tissues. Fetuin-A has been recognized as a multifunctional molecule related to its role in metabolic processes, insulin resistance, regulation of adipogenesis, and mineralization throughout the body. To find out the effect of non-surgical therapy on the periodontal and cardiac parameters and the salivary levels of Vitronectin and Fetuin-A in patients with periodontitis (stage II-III) and coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients within the age group of 30-65 years (male)
3. Patients should have ≥ 10 remaining natural teeth.
4. No history of long term antibiotic use in past 6 months.

Exclusion Criteria:

1. Subjects with systemic conditions such as type I and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies/neoplasm and HIV infection will be excluded from the present investigation.
2. Chronic treatment (>2 weeks) with drugs known to affect periodontal tissues (phenytoin or cyclosporin).
3. Female patients were excluded due to hormonal variations.
4. For Group II and III, subjects on drugs such as corticosteroids, antibiotics, within 6 months of investigation will be excluded.
5. Current smokers and individuals who quit smoking less than 6 months.
6. Patients who have undergone periodontal therapy within the previous 6 months.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male participants are included belonging to 30-65 years of age
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in periodontal parameters | Two years
  Reduction in PPD (measured in mm)
Reduction in periodontal variables | Two years
  Reduction in CAL (measured in mm)
Reduction in periodontal criteria | Two years
  Reduction in Plaque Index (measured in numericals)
Reduction in periodontal variables | Two years
  Reduction in Gingival index (measured in numericals)

CONTACTS AND LOCATIONS:
Locations (1):
- Meenakshi Ammal Dental College and Hospital, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No